CLINICAL TRIAL: NCT03132129
Title: Prevalence and Determinants of Subclinical Cardiovascular Dysfunction in Adults With Type 2 Diabetes Mellitus
Acronym: PREDICT
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0580
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies
Keywords: Type 2 diabetes; Diabetic cardiomyopathy; Cardiovascular magnetic resonance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies | interventions — Diagnostic Imaging; Positron-Emission Tomography; Echocardiography; Exercise Test; Blood Pressure Monitoring, Ambulatory; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Quantitative buffy coat and plasma samples will be stored for future potential biomarker and genotyping studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 diabetics: Participants will be aged (≥18 and ≤75 years) with T2D and no prior history of cardiovascular disease.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance (CMR) imaging and magnetic resonance spectroscopy; Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: Computed tomography coronary artery calcium scoring; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Manganese-enhanced magnetic resonance imaging (MEMRI); Diagnostic Test: Ambulatory blood pressure monitoring; Diagnostic Test: Accelerometer watch; Diagnostic Test: Blood tests
- Healthy controls: Cases will be compared with age-, gender- and ethnicity-matched healthy controls.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance (CMR) imaging and magnetic resonance spectroscopy; Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: Computed tomography coronary artery calcium scoring; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Manganese-enhanced magnetic resonance imaging (MEMRI); Diagnostic Test: Ambulatory blood pressure monitoring; Diagnostic Test: Accelerometer watch; Diagnostic Test: Blood tests

INTERVENTIONS:
Diagnostic Test: Cardiovascular magnetic resonance (CMR) imaging and magnetic resonance spectroscopy — CMR scanning performed on a 3T MRI scanner. Standardised protocol incorporating cine functional assessment to determine LV mass, systolic function and left atrial volumes; global systolic strain and diastolic strain rates will be assessed by tagging and with tissue tracking analysis from cine images, adenosine rest and stress myocardial perfusion to assess reserve index and qualitative perfusion defects as previously described, aortic distensibility and pulse wave velocity to measure aortic stiffness, delayed contrast enhancement for assessment of LV fibrosis and evidence of previous myocardial infarction. Myocardial and liver triglyceride content will be assessed using the modified Hepafat® sequence or 1H MR spectroscopy at the inter ventricular septum. DIXON technique for the quantification of visceral adiposity and subcutaneous adipose tissue.
Diagnostic Test: Transthoracic echocardiography — Comprehensive transthoracic echocardiography, including: tissue Doppler indices of diastolic filling and speckle tracking for systolic and diastolic strain/strain rate, exclusion of valvular abnormalities, assessment of LV size and function.
Diagnostic Test: Computed tomography coronary artery calcium scoring — Computed Tomography coronary calcium scoring to assess the presence of subclinical atherosclerosis and allow an estimate of atheroma burden in addition to epicardial adipose tissue characterisation and systolic strain.
Diagnostic Test: Cardiopulmonary exercise testing — Physician supervised incremental symptom limited cardiopulmonary exercise tolerance test with ECG and haemodynamic monitoring.
Diagnostic Test: Manganese-enhanced magnetic resonance imaging (MEMRI) — A subset of the participants will have cardiac MRI scanning with manganese-based contrast agent, lasting approximately 45-50 minutes. After localisers, baseline functions and native T1 maps have been acquired, Mangafodipir (0.1mL/kg) will be administered intravenously at 1ml/min, with additional T1 maps acquired every 2.5 min after administration of the contrast agent for up to 30 minutes.
Diagnostic Test: Ambulatory blood pressure monitoring — A 24-hour blood pressure monitor will be worn at the end of the visit to the following day.
Diagnostic Test: Accelerometer watch — Watch worn to collect free living physical activity data for 7 days.
Diagnostic Test: Blood tests — Collection of blood samples from each participant to characterise the participant's health status and to develop a proteomic signature of early heart failure.

SUMMARY:
Background: Heart failure is a major cause of morbidity and mortality in diabetes mellitus, but its pathophysiology is poorly understood.

Aim: To determine the prevalence and determinants of subclinical cardiovascular dysfunction in adults with type 2 diabetes (T2D).

Plan: 518 asymptomatic adults (aged 18-75 years) with T2D will undergo comprehensive evaluation of cardiac structure and function using cardiac MRI (CMR) and spectroscopy, echocardiography, CT coronary calcium scoring, exercise tolerance testing and blood sampling. 75 controls will undergo the same evaluation.

Primary hypothesis: myocardial steatosis is an independent predictor of left ventricular global longitudinal strain. Secondary hypotheses: will assess whether CMR is more sensitive to detect early cardiac dysfunction than echocardiography and BNP, and whether cardiac dysfunction is related to peak oxygen consumption.

Expected value of results: This study will reveal the prevalence and determinants of cardiac dysfunction in T2D, and could provide targets for novel therapies.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged ≥18 and ≤75 years.
* Diagnosed with Stable type 2 diabetes (determined by: i) formal diagnosis in GP case records, ii) a record of diagnostic oral glucose tolerance test OR glycated haemoglobin level ≥6.5%).

Exclusion Criteria:

* Angina pectoris or limiting dyspnoea (>NYHA II),
* Major atherosclerotic disease: Symptomatic CAD, history of myocardial infarction, previous revascularisation, stroke/transient ischaemic attack or symptomatic peripheral vascular disease.
* Atrial fibrillation or flutter.
* Moderate or severe valvular heart disease.
* History of heart failure or cardiomyopathy.
* Type 1 diabetes mellitus (T1DM).
* Low fasting C-peptide levels suggestive of adult-onset T1DM.
* Stage III-V renal disease (estimated glomerular filtration rate ≤30ml/min/1.73m2).
* Absolute contraindications to CMR.

Importantly, patients with subclinical CAD, and other common comorbidities such as obesity and hypertension, will not be excluded from this study. This will enable us to evaluate the contribution of CAD to myocardial dysfunction in diabetes and ensures our study group is representative of the general population with diabetes. Similarly, as mild dyspnoea is extremely common and non-specific participants with mild dyspnoea will be included.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases will be adults with stable type 2 diabetes and no past medical history of known cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 593 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of early heart failure in type 2 diabetes | 5 years
  Proportion of participants with type 2 diabetes who have features of early heart failure

SECONDARY OUTCOMES:
Multivariate and independent predictors of LV systolic and diastolic function in type 2 diabetes | 3 years
  Multivariate and independent predictors of LV systolic and diastolic function in type 2 diabetes
Sensitivity of CMR versus echocardiography and BNP for detecting subclinical cardiovascular dysfunction in type 2 diabetes | 3 years
  Sensitivity of CMR versus echocardiography and BNP for detecting subclinical cardiovascular dysfunction in type 2 diabetes
Independent association of CMR measures with aerobic exercise capacity in type 2 diabetes | 3 years
  Independent association of CMR measures (LV systolic and diastolic strain and strain rates) with aerobic exercise capacity (peak VO2) in type 2 diabetes
Differences in LV remodelling (indexed LV mass) between cases and controls | 3 years
  Differences in LV remodelling (indexed LV mass) between cases and controls
Independent clinical and imaging predictors of major adverse cardiovascular and, in particular, heart failure events in the patients with type 2 diabetes | 5 years
  Independent clinical and imaging predictors of major adverse cardiovascular and, in particular, heart failure events in the patients with type 2 diabetes
Differences in cardiac MRI and echo-derived systolic and diastolic strain and strain rates between cases and controls. | 3 years
  Differences in cardiac MRI and echo-derived systolic and diastolic strain and strain rates between cases and controls.
Differences in coronary atheroma burden (CT coronary artery calcium score) between cases and controls | 3 years
  Differences in coronary atheroma burden (CT coronary artery calcium score) between cases and controls
Differences in aerobic exercise capacity (peak V02) between cases and controls | 3 years
  Differences in aerobic exercise capacity (peak V02) between cases and controls
Differences in myocardial perfusion reserve between cases and controls | 3 years
  Differences in myocardial perfusion reserve between cases and controls
Differences in heart rate and blood pressure variability between cases and controls | 3 years
  Differences in heart rate and blood pressure variability between cases and controls
Myocardial steatosis | 3 years
  Myocardial steatosis as an independent predictor of LV global longitudinal strain
Myocardial calcium handling as assessed by manganese-enhanced magnetic resonance imaging (MEMRI) | 5 years
  Manganese influx constants calculated using Patlak modelling
Proteomic signature | 5 years
  Proteomic analysis will be conducted to identify a proteomic signature of early heart failure in type 2 diabetes that will be externally validated
Remission of type 2 diabetes | 5 years
  The phenotype of participants defined as in remission will be compared to active type 2 diabetes and healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Gerry P McCann, MD, Principal Investigator — University of Leicester
Locations (1):
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayton SL, Aslam S, Dattani A, Yeo JL, Gulsin GS, Slomka PJ, Dey D, McCann GP, Singh A. Association of epicardial adipose tissue with markers of cardiac remodelling and clinical outcomes in asymptomatic aortic stenosis. Open Heart. 2026 Feb 9;13(1):e003804. doi: 10.1136/openhrt-2025-003804. PMID 41663151
- [Derived] Yeo JL, Gulsin GS, Brady EM, Dattani A, Bilak JM, Marsh AM, Sian M, Athithan L, Parke KS, Wormleighton J, Graham-Brown MPM, Singh A, Arnold JR, Lawson C, Davies MJ, Xue H, Kellman P, McCann GP. Association of ambulatory blood pressure with coronary microvascular and cardiac dysfunction in asymptomatic type 2 diabetes. Cardiovasc Diabetol. 2022 May 28;21(1):85. doi: 10.1186/s12933-022-01528-2. PMID 35643571